CLINICAL TRIAL: NCT04227899
Title: LIFE-BTK (pivotaL Investigation of saFety and Efficacy of BRS Treatment-Below The Knee) Randomized Controlled Trial
Brief Title: LIFE-BTK Randomized Controlled Trial
Acronym: LIFE-BTK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABT-CIP-10293
Record Dates: First submitted 2020-01-06; First posted 2020-01-14 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Critical Limb Ischemia (CLI)
Keywords: Infrapopliteal lesions; Esprit BTK Everolimus Eluting Bioresorbable Scaffold System; Percutaneous transluminal angioplasty (PTA); ABT-CIP-10293
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Angioplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Esprit BTK (Experimental): Participants who receives Esprit BTK device will be included in this arm
  Interventions: Device: Esprit BTK Device
- Percutaneous Transluminal Angioplasty (PTA) (Active Comparator): Participants who receives PTA treatment will be included in this arm
  Interventions: Device: Percutaneous Transluminal Angioplasty (PTA) Device

INTERVENTIONS:
Device: Esprit BTK Device — Participants will receive Esprit BTK Device
  Arms: Esprit BTK
Device: Percutaneous Transluminal Angioplasty (PTA) Device — Participants will receive PTA treatment
  Arms: Percutaneous Transluminal Angioplasty (PTA)

SUMMARY:
The objective of this prospective, single-blinded, randomized controlled clinical investigation is to evaluate the safety and efficacy of the everolimus eluting Esprit BTK System for the planned treatment of narrowed infrapopliteal lesions. Approximately 225 subjects will be randomized in a 2:1 ratio. The clinical investigation will be conducted at approximately 65 clinical sites in the US, Asia, Australia, and New Zealand.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

1. Subject must provide written informed consent prior to any clinical investigation related procedure.
2. Subject has symptomatic Critical Limb Ischemia (CLI), Rutherford Becker Clinical Category 4 or 5.
3. Subject requires primary treatment of up to two de novo or restenotic (treated with prior PTA) infrapopliteal lesions.
4. Subject must be at least 18 years of age.
5. Female subject of childbearing potential should not be pregnant and must be on birth control.

Note: Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.

Anatomic Inclusion Criteria:

1. Up to two native infrapopliteal lesions, each lesion located in separate infrapopliteal vessel in the same limb. Restenotic (from prior PTA) lesions are allowed.

   1. Lesion must be located in the proximal 2/3 of native infrapopliteal vessels, with vessel diameter of ≥ 2.5 mm and ≤ 4.00 mm by investigator visual assessment.
   2. Total scaffold length to completely cover/treat a target lesion must not exceed 170 mm (total everolimus drug dose of 1790 µg).
   3. The total scaffold length among all target lesions must not exceed 170 mm.
   4. The target vessel cannot have any other angiographic significant lesions (≥50%).
   5. Tandem lesions are allowed if they are < 3 cm apart and the total scaffold length used to cover the entire diseased segment is ≤ 170 mm. Each tandem lesion is considered one lesion.
2. Target lesion(s) must have ≥ 70% stenosis, per visual assessment at the time of the procedure. If needed, quantitative imaging (angiography, IVUS, and/or OCT) can be used to aid accurate sizing of the vessels.
3. The distal margin of the target lesion must be located ≥ 10 cm proximal to the proximal margin of the ankle mortise. The vessel segment distal to the target lesion must be patent all the way to the ankle, with no significant lesion (≥ 50% stenosis).
4. Significant lesion (≥ 50% stenosis) in the inflow artery(ies) must be treated successfully (as per physician's assessment of the angiography) through standard of care prior to the treatment of the target lesion. Treatment can be done within the same trial procedure.
5. Non-target lesion(s) (if applicable) must be located in separate infrapopliteal vessel(s) from the target lesion, and suitable to be treated per institution standard of care.
6. Guidewire must cross the target lesion successfully. Crossing in an antegrade fashion is preferred, but retrograde crossing may be used. However, the treatment must be delivered antegrade.

Exclusion Criteria:

General Exclusion Criteria:

1. Subject is currently participating in another clinical investigation that has not yet completed its primary endpoint.
2. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period.
3. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements.
4. Incapacitated individuals, defined as persons who are mentally ill, mentally handicapped, or individuals without legal authority, are excluded from the study population.
5. Subject has had any amputation to the ipsilateral extremity other than the toe or forefoot, or subject has had major amputation to the contralateral extremity < 1 year prior to index procedure and is not independently ambulating.
6. Subject has known hypersensitivity or contraindication to device material and its degradants (everolimus, poly (L-lactide), poly (DL-lactide), lactide, lactic acid) and cobalt, chromium, nickel, platinum, tungsten, acrylic and fluoro polymers that cannot be adequately pre-medicated. Subject has a known contrast sensitivity that cannot be adequately pre-medicated.
7. Subject has known allergic reaction, hypersensitivity or contraindication to aspirin; or to ADP antagonists such clopidogrel, prasugrel or ticagrelor; or to anticoagulants such as heparin or bivalirudin, and therefore cannot be adequately treated with study medications. Subject with planned surgery or procedure necessitating discontinuation of antiplatelet medications, within 12 months after index procedure. Planned amputation that will necessitate discontinuation of antiplatelet medications is allowed.
8. Subject has life expectancy ≤ 1 year.
9. Subject has had a stroke within the previous 3 months with residual Rankin score of ≥ 2.
10. Subject has renal insufficiency as defined as an estimated GFR < 30 ml/min per 1.73m^2.
11. Subject is currently on dialysis.
12. Subject has platelet count < 100,000 cells/mm^3 or > 700,000 cells/mm^3, a WBC < 3,000 cells/mm^3, or hemoglobin < 9.0 g/dl.
13. Subject has known serious immunosuppressive disease (e.g., human immunodeficiency virus), or has severe autoimmune disease, that requires chronic immunosuppressive therapy (e.g., systemic lupus erythematosus, etc.), or subject is receiving immunosuppression therapy for other conditions. Subjects treated for HIV (Human Immunodeficiency Virus) and who have undetectable viral load, such that their immune system is not considered compromised, are eligible.
14. Subject has Body Mass Index (BMI) <18.
15. Subject is receiving or scheduled to receive anticancer therapy for malignancy within 6 months prior to index procedure or within 1 year after the procedure. Patients taking medications classified as chemotherapy but who have been in remission for at least 6 months are eligible.
16. Subject has coagulation disorder that increases the risk of arterial thrombosis. Subjects with deep vein thrombosis and disorders that increase the risk of deep vein thrombosis can be included in the study.
17. Subject who requires thrombolysis as a primary treatment modality or requires other treatment for acute limb ischemia of the target limb.
18. Subject has previously had, or requires surgical revascularization involving any vessel of the ipsilateral extremity. Prior femoropopliteal or aortobifemoral bypass is allowed. Any bypass to the tibial arteries is not allowed.
19. Subject has signs or symptoms of advanced limb infection or septicemia (fever > 38.5, WBC > 15,000 cells/microliter, hypotension) at the time of assessment. Osteomyelitis of the phalanges or metatarsal heads (as described in exclusion criteria #21a) or cellulitis of the foot amenable to treatment with IV antibiotics at the time of revascularization is acceptable.
20. Subject is bedridden or unable to walk (with assistance is acceptable). Subjects in wheelchair who are able to mobilize on their own can be enrolled.
21. Subject with extensive tissue loss salvageable only with complex foot reconstruction or non-traditional transmetatarsal amputations. This includes subjects with:

    1. Osteomyelitis that extends proximal to the metatarsal heads. Osteomyelitis limited to the phalanges or metatarsal heads is acceptable for enrollment.
    2. Gangrene involving the plantar skin of the forefoot, midfoot, or heel.
    3. Deep ulcer or large shallow ulcer (> 3 cm) involving the plantar skin of the forefoot, midfoot, or heel.
    4. Full thickness heel ulcer with/without calcaneal involvement.
    5. Any wound with calcaneal bone involvement.
    6. Wounds that are deemed to be neuropathic or non-ischemic in nature.
    7. Wounds that would require flap coverage or complex wound management for large soft tissue defect.
    8. Full thickness wounds on the dorsum of the foot with exposed tendon or bone.
22. Subject is unable or unwilling to provide written consent prior to enrollment.
23. Subject has active symptoms and/or a positive test result of COVID-19 or other rapidly spreading novel infectious agent within the prior 2 months.

Anatomic Exclusion Criteria:

1. Lesions with severe calcification, in which there is a high likelihood that successful pre-dilatation cannot be achieved.
2. Lesion that has prior metallic stent implant.
3. Significant (≥ 50% stenosis) lesion in a distal outflow artery that would be perfused by the target vessel and that requires treatment at the time of the index procedure.
4. Subject has had or will require treatment in any vessel with an everolimus drug-coated or drug-eluting device < 30 days pre-study procedure, or during the index procedure, such that the cumulative (Esprit BTK plus everolimus-eluting device) everolimus drug dose exceeds 1790 μg.
5. Target or (if applicable) non-target vessel contains visible thrombus as indicated in the angiographic images.
6. Subject has angiographic evidence of thromboembolism or atheroembolism in the ipsilateral extremity. (Pre- and post-angiographic imaging must confirm the absence of emboli in the distal anatomy).
7. Unsuccessfully treated proximal inflow limiting arterial stenosis or inflow-limiting arterial lesions left untreated.
8. No angiographic evidence of a patent pedal artery.
9. Target or (if applicable) non-target lesion location requiring bifurcation treatment method that requires scaffolding of both branches (provisional treatment, without intention of scaffolding both branches is acceptable).
10. Aneurysm in the iliac, common femoral, superficial femoral, popliteal or target artery of the ipsilateral extremity.
11. Visual assessment of the target lesion suggests that the investigator is unable to pre-dilate the lesion according to the vessel diameter.
12. Target lesion has a high probability that atherectomy will be required at the time of index procedure for treatment of the target vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2027-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ramon L Varcoe, MBBS, MS, FRACS, PhD, Principal Investigator — Prince of Wales Private Hospital, Randwick, NSW, Australia; Sahil Parikh, MD, FACC, FSCAI, Principal Investigator — New York Presbyterian Hospital, New York, NY; Brian DeRubertis, MD, FACS, Principal Investigator — NewYork-Presbyterian/Weill Cornell Medical Center, New York, NY
Locations (50):
- United States (43):
  - Comprehensive Integrated Care, Gilbert, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - St. Helena Hospital, Deer Park, California
  - Mission Cardiovascular Research Institute, Fremont, California
  - UCSF Fresno, Fresno, California
  - St. Joseph Hospital, Orange, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Manatee Memorial Hospital, Bradenton, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Palm Vascular Centers, Miami Beach, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - The Iowa Clinic, West Des Moines, Iowa
  - Via Christi Regional Medical Center - St. Francis Campus, Wichita, Kansas
  - Cardiovascular Institute of the South, Houma, Louisiana
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Charlton Memorial Hospital, Russells Mills, Massachusetts
  - Jackson Heart Clinic, Jackson, Mississippi
  - Deborah Heart & Lung Center, Browns Mills, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Vascular Institute of Atlantic Medical Imaging, Pomona, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - NYU Langone Health, New York, New York
  - Mount Sinai Hospital, New York, New York
  - New York-Presbyterian/Columbia University Medical Center, New York, New York
  - New York Presbyterian Hospital/Cornell University, New York, New York
  - James J. Peters VA Medical Center, The Bronx, New York
  - NC Heart & Vascular Research, Raleigh, North Carolina
  - The Lindner Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ascension St. John Jane Phillips, Bartlesville, Oklahoma
  - Lankenau Institute for Medical Research, Bryn Mawr, Pennsylvania
  - Saint Vincent Consultants in Cardiovascular Diseases, Erie, Pennsylvania
  - Pinnacle Health System, Wormleysburg, Pennsylvania
  - Anmed Health, Anderson, South Carolina
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - Texas Tech University Health Sciences Center at Lubbock, Lubbock, Texas
  - San Antonio Vascular and Endovascular Clinic, San Antonio, Texas
- Australia (2):
  - Prince of Wales Private Hospital, Randwick, New South Wales
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Auckland City Hospital, Auckland, Auckland, New Zealand
- Changi General Hospital, Singapore, Singapore
- National Taiwan University Hospital, Taipei, Zhongzheng, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeRubertis BG, Varcoe RL, Krishnan P, Bonaca MP, O'Connor DJ, Pin R, Metzger DC, Holden A, Lee JK, Iida O, Armstrong EJ, Kum SWC, Kolluri R, Bajakian DR, Garcia LA, Shishehbor MH, Yu S, Ruster K, Martinsen BJ, Igyarto Z, Parikh SA. Drug-Eluting Resorbable Scaffold Versus Balloon Angioplasty for Below-the-Knee Peripheral Artery Disease: 2-Year Results From the LIFE-BTK Trial. Circulation. 2025 Oct 14;152(15):1076-1086. doi: 10.1161/CIRCULATIONAHA.125.075080. Epub 2025 Sep 10. PMID 40927852
- [Derived] Varcoe RL, DeRubertis BG, Kolluri R, Krishnan P, Metzger DC, Bonaca MP, Shishehbor MH, Holden AH, Bajakian DR, Garcia LA, Kum SWC, Rundback J, Armstrong E, Lee JK, Khatib Y, Weinberg I, Garcia-Garcia HM, Ruster K, Teraphongphom NT, Zheng Y, Wang J, Jones-McMeans JM, Parikh SA; LIFE-BTK Investigators. Drug-Eluting Resorbable Scaffold versus Angioplasty for Infrapopliteal Artery Disease. N Engl J Med. 2024 Jan 4;390(1):9-19. doi: 10.1056/NEJMoa2305637. Epub 2023 Oct 25. PMID 37888915

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 261 subjects from 50 sites were registered in the RCT population of the study including 88 in the PTA group and 173 in the Esprit BTK group up to 1-year follow-up, between August 18, 2020, and September 14, 2022.
Groups:
- Esprit BTK: Participants who receive Esprit BTK device will be included in this arm
  Esprit BTK Device: Participants will receive Esprit BTK Device
- Percutaneous Transluminal Angioplasty (PTA): Participants who receive PTA treatment will be included in this arm
  Percutaneous Transluminal Angioplasty (PTA) Device: Participants will receive PTA treatment
Period: Overall Study
Arm/Group | Esprit BTK | Percutaneous Transluminal Angioplasty (PTA)
Started | 173 | 88
Completed | 153 | 78
Not Completed | 20 | 10
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Death | 12 | 6
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esprit BTK | Percutaneous Transluminal Angioplasty (PTA) | Total
Number analyzed (Participants) | 173 | 88 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (9.9) | 71.1 (10.4) | 72.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 27 | 83
  Male | 117 | 61 | 178
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 12 | 43
  Not Hispanic or Latino | 132 | 70 | 202
  Unknown or Not Reported | 10 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 36 | 11 | 47
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 21 | 11 | 32
  White | 97 | 56 | 153
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 18 | 7 | 25
Hypertension [Count of Participants; unit: Participants] | 163 | 80 | 243

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: Number of Participants With Composite of Limb Salvage and Primary Patency
Description: This endpoint was to evaluate the effectiveness of the Esprit BTK System in maintaining patency (CD-TLR and binary restenosis), and at preventing catastrophic limb events such as total vessel occlusion or major amputation. Composite of Limb Salvage and Primary Patency included freedom from: above ankle amputation in index limb, 100% total occlusion of target vessel, binary restenosis of target lesion and clinically-driven target lesion revascularization (CD-TLR).
Time Frame: At 1 year
Population: Analysis excluded subjects who terminated from the study prior to the lower limit (337 days) of the 1-year primary efficacy endpoint follow-up window without any components of the primary endpoint, and subjects with no known endpoint event and who did not have analyzable duplex ultrasound or angiography for the 1-year imaging assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Esprit BTK | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 149 | 71
Participants | 111 | 31
Statistical Analysis 1: Comparison: Esprit BTK vs Percutaneous Transluminal Angioplasty (PTA); Test type: Other; p < 0.0001, One-sided Chi-square test

2. Primary Outcome: Primary Safety Endpoint: Freedom From Major Adverse Limb Event + Peri-Operative Death Rate (MALE + POD)
Description: The primary safety endpoint assessed the safety of the devices used for treatment of below the knee lesions. It included freedom from MALE+POD (Major Adverse Limb Event + Peri-Operative Death). MALE includes above-ankle amputation in the index limb, major re-intervention on the index limb at 6 months and POD includes perioperative (30-day) mortality.
Time Frame: At 30 days (for POD) and 6 months (for MALE)
Population: Analysis excluded subjects who terminated from the study prior to the lower limit (152 days) of the 6-month primary safety endpoint follow-up window without any components of the primary endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Esprit BTK | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 160 | 85
Participants | 155 | 85
Statistical Analysis 1: Comparison: Esprit BTK vs Percutaneous Transluminal Angioplasty (PTA); Test type: Other; p = 0.0019, Farrington-Manning non-inferiority (NI)

3. Secondary Outcome: First Powered Secondary Endpoint: Binary Restenosis of the Target Lesion
Description: This endpoint was added to better evaluate the device performance as binary restenosis was used as a marker for disease progression over time.
Time Frame: At 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Esprit BTK | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 149 | 71
Participants | 35 | 35
Statistical Analysis 1: Comparison: Esprit BTK vs Percutaneous Transluminal Angioplasty (PTA); Test type: Other; p < 0.0001, Chi-squared

4. Secondary Outcome: Second Powered Secondary Endpoint: Freedom From Above Ankle Amputation in Index Limb, 100% Total Occlusion of the Target Vessel, and CD-TLR.
Description: This endpoint was chosen as it was important to assess whether Esprit BTK System was efficacious at maintaining patency and preventing catastrophic limb events through 1 year.
Time Frame: At 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Esprit BTK | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 149 | 71
Participants | 124 | 49
Statistical Analysis 1: Comparison: Esprit BTK vs Percutaneous Transluminal Angioplasty (PTA); Test type: Other; p = 0.0081, One-sided Chi-square test

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Esprit BTK | Percutaneous Transluminal Angioplasty (PTA)
All-Cause Mortality (participants affected / at risk) | 12/173 | 6/88
Serious Adverse Events (participants affected / at risk) | 89/173 | 45/88
Other Adverse Events (participants affected / at risk) | 105/173 | 60/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esprit BTK (N=173) | Percutaneous Transluminal Angioplasty (PTA) (N=88)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 3
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 | 0
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0
AORTIC VALVE STENOSIS (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 4 | 2
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 1 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 5 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 2 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 | 0
CYANOSIS (Cardiac disorders) | 1 | 0
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 4 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
MELAENA (Gastrointestinal disorders) | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
ASTHENIA (General disorders) | 2 | 1
CHEST PAIN (General disorders) | 2 | 1
DEATH (General disorders) | 6 | 0
OEDEMA PERIPHERAL (General disorders) | 2 | 0
PYREXIA (General disorders) | 0 | 1
ULCER (General disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 0
CELLULITIS (Infections and infestations) | 5 | 2
CORONA VIRUS INFECTION (Infections and infestations) | 2 | 1
DIABETIC FOOT INFECTION (Infections and infestations) | 1 | 0
GANGRENE (Infections and infestations) | 4 | 2
IMPLANT SITE INFECTION (Infections and infestations) | 1 | 0
INCISION SITE ABSCESS (Infections and infestations) | 1 | 0
INCISION SITE INFECTION (Infections and infestations) | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 2 | 1
OSTEOMYELITIS CHRONIC (Infections and infestations) | 1 | 0
PAROTITIS (Infections and infestations) | 1 | 0
PERIRECTAL ABSCESS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 3 | 3
POST PROCEDURAL INFECTION (Infections and infestations) | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 0 | 1
RHINOVIRUS INFECTION (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 2 | 1
SEPTIC SHOCK (Infections and infestations) | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 2 | 0
WOUND INFECTION (Infections and infestations) | 1 | 0
ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 9 | 7
FALL (Injury, poisoning and procedural complications) | 6 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
SKIN WOUND (Injury, poisoning and procedural complications) | 7 | 2
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
TENDON INJURY (Injury, poisoning and procedural complications) | 0 | 1
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 2 | 0
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 15 | 5
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 1
ANTICOAGULATION DRUG LEVEL BELOW THERAPEUTIC (Investigations) | 0 | 1
DEVICE FUNCTION TEST (Investigations) | 1 | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 1
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 0 | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 9 | 4
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
APHASIA (Nervous system disorders) | 0 | 1
CAROTID ARTERY DISEASE (Nervous system disorders) | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 | 0
COGNITIVE DISORDER (Nervous system disorders) | 1 | 1
CONVULSION (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 1
MYELOPATHY (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 2 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1
DELIRIUM (Psychiatric disorders) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 4 | 2
RENAL FAILURE ACUTE (Renal and urinary disorders) | 6 | 2
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 | 0
DYSPNOEA PAROXYSMAL NOCTURNAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 7 | 1
CARDIAC PACEMAKER INSERTION (Surgical and medical procedures) | 0 | 1
FOOT AMPUTATION (Surgical and medical procedures) | 2 | 0
OSTEOTOMY (Surgical and medical procedures) | 1 | 0
PERIPHERAL REVASCULARISATION (Surgical and medical procedures) | 4 | 1
TOE AMPUTATION (Surgical and medical procedures) | 8 | 4
VASCULAR STENT INSERTION (Surgical and medical procedures) | 1 | 0
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 7 | 2
ARTERIAL RUPTURE (Vascular disorders) | 1 | 0
ARTERIAL STENOSIS (Vascular disorders) | 1 | 0
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 2 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
EMBOLISM (Vascular disorders) | 1 | 0
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 1 | 0
HAEMATOMA (Vascular disorders) | 1 | 0
HAEMORRHAGE (Vascular disorders) | 5 | 2
HYPERTENSION (Vascular disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 2 | 0
INTERMITTENT CLAUDICATION (Vascular disorders) | 0 | 1
PERIPHERAL ARTERY DISSECTION (Vascular disorders) | 0 | 2
PERIPHERAL EMBOLISM (Vascular disorders) | 1 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 2 | 1
THROMBOSIS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esprit BTK (N=173) | Percutaneous Transluminal Angioplasty (PTA) (N=88)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
ANGINA UNSTABLE (Cardiac disorders) | 1 | 1
ARRHYTHMIA (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 4 | 1
BRADYCARDIA (Cardiac disorders) | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 1 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0
DEAFNESS (Ear and labyrinth disorders) | 1 | 0
EAR HAEMORRHAGE (Ear and labyrinth disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0
HYPOTHYROIDISM (Endocrine disorders) | 1 | 0
CATARACT (Eye disorders) | 0 | 1
VISION BLURRED (Eye disorders) | 1 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 0
COLONIC POLYP (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
ASTHENIA (General disorders) | 1 | 1
CHEST PAIN (General disorders) | 2 | 4
CHILLS (General disorders) | 1 | 0
FATIGUE (General disorders) | 1 | 0
HYPOTHERMIA (General disorders) | 0 | 1
OEDEMA (General disorders) | 2 | 0
OEDEMA PERIPHERAL (General disorders) | 5 | 2
PYREXIA (General disorders) | 2 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 | 0
HEPATITIS (Hepatobiliary disorders) | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 0 | 1
BRONCHITIS (Infections and infestations) | 1 | 0
CELLULITIS (Infections and infestations) | 4 | 1
CORONA VIRUS INFECTION (Infections and infestations) | 4 | 4
FUNGAL SKIN INFECTION (Infections and infestations) | 0 | 1
GANGRENE (Infections and infestations) | 1 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 0
PARONYCHIA (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 1 | 1
TINEA VERSICOLOUR (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 3 | 0
WOUND INFECTION (Infections and infestations) | 1 | 1
ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 5 | 4
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0
EYELID INJURY (Injury, poisoning and procedural complications) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 3 | 4
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
INCISION SITE HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
INCISION SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 1
OPEN WOUND (Injury, poisoning and procedural complications) | 0 | 1
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SKIN WOUND (Injury, poisoning and procedural complications) | 11 | 7
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
TENDON INJURY (Injury, poisoning and procedural complications) | 0 | 1
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 2 | 1
WOUND (Injury, poisoning and procedural complications) | 2 | 0
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 10 | 6
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 2 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 0
BLOOD PRESSURE INCREASED (Investigations) | 1 | 0
CORONAVIRUS TEST POSITIVE (Investigations) | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1
OXYGEN SATURATION DECREASED (Investigations) | 1 | 0
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 1 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 | 0
GOUT (Metabolism and nutrition disorders) | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
NUCHAL RIGIDITY (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 21 | 15
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
ABDOMINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ADRENAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ATAXIA (Nervous system disorders) | 1 | 0
CAROTID ARTERY DISEASE (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
COGNITIVE DISORDER (Nervous system disorders) | 1 | 0
COMA (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 2 | 1
HYPOAESTHESIA (Nervous system disorders) | 1 | 1
INTRAVENTRICULAR HAEMORRHAGE (Nervous system disorders) | 1 | 0
POLYNEUROPATHY (Nervous system disorders) | 2 | 1
PRESYNCOPE (Nervous system disorders) | 1 | 1
SCIATICA (Nervous system disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0
DELIRIUM (Psychiatric disorders) | 0 | 1
DYSURIA (Renal and urinary disorders) | 1 | 0
PYURIA (Renal and urinary disorders) | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 5 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BLISTER (Skin and subcutaneous tissue disorders) | 1 | 0
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 | 2
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 1
SCAB (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN SWELLING (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 3 | 0
AMNIOTIC MEMBRANE GRAFT (Surgical and medical procedures) | 1 | 0
CARDIAC ABLATION (Surgical and medical procedures) | 0 | 1
FOOT AMPUTATION (Surgical and medical procedures) | 1 | 0
INCISIONAL HERNIA REPAIR (Surgical and medical procedures) | 1 | 0
PERIPHERAL REVASCULARISATION (Surgical and medical procedures) | 0 | 4
REMOVAL OF FOREIGN BODY (Surgical and medical procedures) | 0 | 1
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 11 | 3
ARTERIAL RUPTURE (Vascular disorders) | 3 | 0
ARTERIAL STENOSIS (Vascular disorders) | 0 | 1
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 1 | 0
ARTERY DISSECTION (Vascular disorders) | 1 | 0
EMBOLISM (Vascular disorders) | 0 | 1
HAEMATOMA (Vascular disorders) | 4 | 0
HAEMORRHAGE (Vascular disorders) | 3 | 1
HYPERTENSION (Vascular disorders) | 4 | 1
HYPOTENSION (Vascular disorders) | 2 | 0
ILIAC ARTERY STENOSIS (Vascular disorders) | 0 | 1
INTERMITTENT CLAUDICATION (Vascular disorders) | 0 | 2
LABILE BLOOD PRESSURE (Vascular disorders) | 1 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 1
PERIPHERAL ARTERY DISSECTION (Vascular disorders) | 2 | 3
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 1
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 1 | 0
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 0 | 1
VASOSPASM (Vascular disorders) | 1 | 0
VENOUS INSUFFICIENCY (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT04227899/Prot_002.pdf
  • Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT04227899/SAP_003.pdf